CLINICAL TRIAL: NCT01252615
Title: Patient and Intimate Partner Intervention to Improve Outcomes After an ICD
Brief Title: Patient and Partner Intervention After an Implantable Cardioverter Defibrillator (ICD)
Acronym: P+P
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Cynthia M. Dougherty, Professor, Biobehavioral Nursing and Health Systems, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36576-C
Record Dates: First submitted 2010-11-18; First posted 2010-12-03 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Implantable Cardioverter Defibrillator (ICD)
Keywords: ICD; HF; cardiac arrest; VF; cardiac arrhythmias
MeSH Terms: conditions — Heart Arrest; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient only (Experimental): Patient with the ICD is involved in the intervention
  Interventions: Behavioral: patient only
- patient and partner (Experimental): patient with the ICD and intimate partner are involved in the intervention
  Interventions: Behavioral: patient and partner intervention

INTERVENTIONS:
Behavioral: patient only — education, behavioral strategies, psychological interventions
  Arms: patient only
Behavioral: patient and partner intervention — education, psychological support, behavioral strategies
  Arms: patient and partner

SUMMARY:
The goal of this study is to compare a patient only to a patient+partner intervention on recovery outcomes of patients and partners after Implantable Cardioverter Defibrillator (ICD) implantation.

DETAILED DESCRIPTION:
The goal of this randomized trial is to test a patient+partner intervention against the patient only intervention on recovery outcomes of patients and partners after ICD implantation. By interventing with both ICD patients and their partners, we expect to further improve outcomes of patients and aid in recovery of partners. Over a five year period we will test the effects of a 12 week patient+partner intervention against a patient only intervention in the first year subsequent to ICD implantation, using a 2 group (N=150/group) randomized clinical trial design. Relevant data will be collected on ICD patients and intimate partners at hospital discharge, 1, 3, 6, 12 months post-ICD implantation. The four major outcomes are: physical functioning, psychological adjustment, health care utilization, and relationship impact. The primary analysis of treatment effect is the change in outcome variables from baseline to 3 months for the patient and partner. Secondarily, exploring long term effects of the intervention, theoretical elements, and the intervention effects by ICD implant reason will be determined.

ELIGIBILITY:
Inclusion Criteria:

* first ICD implantation due to either primary or secondary prevention of SCA
* intimate partner (spouse, lover, or life partner) living at the same residence and willing to participate
* able to read, speak, and write English
* access to telephone for 1 year after ICD implantation

Exclusion Criteria:

* clinical co-morbidities that severely impair cognitive and physical functioning at telephone screening
* Short BLESSED score > 6
* age less than 21 years
* AUDIT-C score > 4 for alcohol use
* ASSIST 2.0 score > 4 for daily non-medical use of opiates or hallucinogens,

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2009-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Physical functioning | 3 months
  symptoms, health related quality of life, steps/day

SECONDARY OUTCOMES:
psychological adjustment | 3 months
  anxiety, depression, ICD acceptance

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Dougherty, PhD, Principal Investigator — University of Washington
Locations (1):
- Cynthia M. Dougherty, Seattle, Washington, United States

REFERENCES:
- [Derived] Liberato ACS, Thompson EA, Dougherty CM. Intervention mediating effects of self-efficacy on patient physical and psychological health following ICD implantation. J Behav Med. 2021 Dec;44(6):842-852. doi: 10.1007/s10865-021-00244-8. Epub 2021 Jul 23. PMID 34302228
- [Derived] Dougherty CM, Thompson EA, Kudenchuk PJ. Patient plus partner trial: A randomized controlled trial of 2 interventions to improve outcomes after an initial implantable cardioverter-defibrillator. Heart Rhythm. 2019 Mar;16(3):453-459. doi: 10.1016/j.hrthm.2018.10.011. Epub 2018 Oct 16. PMID 30340060
- [Derived] Lau ET, Thompson EA, Burr RL, Dougherty CM. Safety and Efficacy of an Early Home-Based Walking Program After Receipt of an Initial Implantable Cardioverter-Defibrillator. Arch Phys Med Rehabil. 2016 Aug;97(8):1228-36. doi: 10.1016/j.apmr.2016.02.007. Epub 2016 Mar 3. PMID 26940383
- [Derived] Dougherty CM, Thompson EA, Kudenchuk PJ. Development and testing of an intervention to improve outcomes for partners following receipt of an implantable cardioverter defibrillator in the patient. ANS Adv Nurs Sci. 2012 Oct-Dec;35(4):359-77. doi: 10.1097/ANS.0b013e318271d2e8. PMID 23107992